CLINICAL TRIAL: NCT00758732
Title: A Multicenter Randomized Phase II Study of Docetaxel/Carboplatin Versus Docetaxel/Pegylated Liposomal Doxorubicin as Second Line Treatment in Patients With Platinum Sensitive Disease
Brief Title: Docetaxel/Carboplatin Versus Docetaxel/Caelyx in Pretreated Patients With Ovarian Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/05.09
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Ovarian Cancer
Keywords: Cancer; Ovarian cancer; Chemotherapy; Docetaxel; Carboplatin; Pegylated doxorubicin; Platinum sensitive
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Docetaxel; Carboplatin; liposomal doxorubicin

ARMS (2):
- 1 (Experimental): Docetaxel/carboplatin
  Interventions: Drug: Docetaxel; Drug: Carboplatin
- 2 (Experimental): Docetaxel/Caelyx
  Interventions: Drug: Docetaxel; Drug: Liposomal doxorubicin

INTERVENTIONS:
Drug: Docetaxel — Docetaxel at the dose of 75mg/m2 over a 60 min intravenous infusion every 3 weeks for a maximum of 6 consecutive cycles
  Other Names: Taxotere
  Arms: 1
Drug: Carboplatin — Carboplatin 5 AUC over a 90 min intravenous infusion every 3 weeks for a maximum of 6 consecutive cycles
  Arms: 1
Drug: Docetaxel — Docetaxel at the dose of 40mg/m2 over a 60 min intravenous infusion every 2 weeks in 28 days cycle for a maximum of 6 consecutive cycles.
  Other Names: Taxotere
  Arms: 2
Drug: Liposomal doxorubicin — Liposomal doxorubicin at the dose of 20 mg/m2 over a 90 min intravenous infusion every 2 weeks in 28 days cycle for a maximum of 6 consecutive cycles.
  Other Names: Caelyx
  Arms: 2

SUMMARY:
This trial will compare the efficacy of docetaxel/carboplatin versus docetaxel/liposomal doxorubicin in pretreated patients with advanced ovarian carcinoma and treatment free-interval of at least six months

DETAILED DESCRIPTION:
The second-line treatment in advanced ovarian cancer has been proved effective in prolonging overall survival and improving quality of life. In patients with platinum-sensitive ovarian cancer (relapsed disease after 6 months from the end of first line chemotherapy) the combination of paclitaxel/carboplatin is considered the standard treatment. Generally, the combination platinum-based chemotherapy may well be associated with a survival benefit in patients with platinum-sensitive disease. Carboplatin, pegylated doxorubicin (caelyx) docetaxel, have been approved for second-line treatment of ovarian carcinoma and seem to be active in platinum-sensitive disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian cancer
* Stage IIIB/IV
* Failure to prior chemotherapy with paclitaxel /carboplatin regimen and treatment free interval > 6 months
* Presence of two-dimensional measurable disease.
* Life expectancy of more than 3 months.
* Age ≥ 18 years.
* Performance status (WHO) 0-2
* Adequate bone marrow function (Absolute neutrophil count >1000/mm^3, Platelet count>100000/mm^3, Hemoglobin>9gr/mm^3)
* Adequate liver (Bilirubin<1.5 times upper limit of normal and SGOT/SGPT<2 times upper limit of normal) and renal function (creatinine<2mg/dl)
* Informed consent

Exclusion Criteria:

* Pregnant or nursing
* Psychiatric illness or social situation that would preclude study compliance'
* Other concurrent uncontrolled illness
* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Toxicity profile | Toxicity assessment on each cycle
Time to tumor progression | 1 year
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christos Emmanouilides, MD, Principal Investigator — Interbalkan Hospital, division of Oncology, Pylaia, Thessaloniki
Locations (12):
- Greece (12):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athnes, Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - Department of Medical Oncology, "Marika Iliadis" Hospital of Athens, Athens
  - Department of Medical Oncology, Air Forces Military Hospital of Athens, Athens
  - Medical Oncology Unit, 401 Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - First Department of Medical Oncology, "Metaxa's" Anticancer Hospital of Pireas, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki
  - Interbalkan Hospital, division of Oncology, Pylaia, Thessaloniki, Thessaloniki
  - Medical Oncology Unit, "AXEPA" General Hospital of Thessaloniki, Thessaloniki